CLINICAL TRIAL: NCT05444660
Title: A Retrospective Post Market Clinical Follow-up (PMCF) Study Evaluating the Safety and Clinical Performance of the SABER (OTW) PTA Dilatation Catheter, SABERX PTA Dilatation Catheter, and Powerflex Pro PTA Catheter Used in Infra-popliteal Vessels, During Percutaneous Transluminal Angioplasty (PTA) Procedures.
Brief Title: PMCF Study for Peripheral Arteries Below the Knee (BTK)
Status: Completed | Type: Observational
Sponsor: Cordis US Corp. (Industry)
Collaborators: FCRE (Foundation for Cardiovascular Research and Education) (Other)
Responsible Party: Sponsor
Other Study IDs: FCRE 220104
Record Dates: First submitted 2022-04-14; First posted 2022-07-06 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The rationale of this study is to confirm and support the clinical safety and performance of any of these products in a real-word population of 100 patients who underwent an endovascular intervention within standard-of-care (SOC) of the infra-popliteal vessels, using at least one of the products (named above) from Cordis US Corp.

DETAILED DESCRIPTION:
Peripheral artery disease can be a severe and complex condition that is still a challenge for both surgical and endovascular therapies (1,2). Arterial disease is known to be located predominantly in the superficial femoral artery in patients with claudication and in the below-the-knee (BTK) region in patients with critical limb ischemia (CLI). Especially in patients with diabetes (3-5), -where arterial disease is commonly characterized by long, multilevel disease involving all infrapopliteal vessels-the risk of peripheral artery disease is significantly higher and tends to be more aggressive than in patients without diabetes.

Infrapopliteal arterial occlusive disease afflicts numerous patients with pain at rest, ischemic ulceration, or gangrene (6-7). Critical limb ischemia (CLI) mainly results from this disease. In general, patients suffering from CLI have many comorbidities, such as diabetes mellitus and end-stage renal disease, and often have high morbidity, mortality, and consumption of health care and social care resources (6). Therefore, effectual management is urgently required for patients with CLI.

With the rapid improvements in endovascular instruments and experience of physicians, endovascular therapy has become a major option for the revascularization of infrapopliteal occlusive arteries. Percutaneous transluminal angioplasty (PTA) is the most commonly used endovascular therapy for this disease, especially during the initial onset of CLI. Currently, PTA is considered an effective treatment because of its minimal invasiveness, shortened hospitalization time, and acceptable patency rate (8-9). In recent years, several studies have assessed the safety and efficacy of PTA.

In this regard, the purpose of the current post market clinical follow-up (PMCF) trial is to assess the safety and efficacy of different CE-marked medical devices from Cordis (SABER OTW PTA Dilatation Catheter, SABERX PTA Dilatation Catheter, and Powerflex Pro PTA Catheter) used in the infrapopliteal vessels BTK, when used as intended by the manufacturer (i.e., adhering to the Instruction for Use - IFU). The devices under investigation in the current study are the SABER OTW PTA Dilatation Catheter, SABERX PTA Dilatation Catheter, and Powerflex Pro PTA Catheter, which are described in detail in section 3.1.

Also, data will be collected which may also include acute outcomes for the additional supportive devices listed below in detail in section 4. that may have been used during peripheral angioplasty procedure. However, these devices are not a part of the study devices and would not affect the inclusion criteria for study. The additional devices include the Cordis guidewires (Emerald, ATW, Stablizer, Storq, SV 0.018", Wizdom), Cordis guiding catheters (Adroit, Vista Brite Tip), Cordis diagnostic catheters (Super Torque, Super Torque MB, Super Torque Plus, Infiniti 4F/5F/6F, Tempo 4F, Tempo Aqua, High Flow, Pigtail Straightener), Cordis vascular access devices (Avanti+, Brite Tip, Vista Brite IG, vessel dilator), Cordis vascular closure devices (MynxGrip and Mynx Control) and Cordis OUTBACK CTO catheters which may be used during peripheral angioplasty procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is >18 years old.
2. Target Lesion is located in the infrapopliteal arteries.
3. Patient who underwent treatment (PTA) in the infrapopliteal vessels with at least one of the SABER OTW PTA Catheter the SABERX PTA Catheter and/or the Powerflex Pro PTA Catheter as described in the IFU for each device.

Exclusion Criteria:

1. Anatomy or size of vessels that would have not allowed appropriate usage of the study devices, following IFU of the study devices.
2. Patients who were not suitable for receiving interventional surgeries of lower limb arteries for treatment.
3. Women who were pregnant or lactating at time of the procedure.
4. Any patient who was considered to be hemodynamically unstable at onset of procedure.
5. Patient was not available for follow up at the clinical site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diseased patients with PAD who underwent an endovascular intervention within standard-of-care (SOC) of the infra-popliteal vessels. In this PMCF study, data from minimally invasive medical devices will be collected. Indications for which the study devices are intended are listed in section 3.1. Patient's data will be selected based on the investigator's assessment and evaluation of the underlying disease. The patient's medical condition should have been stable, with no underlying medical condition which would prevent them from undergoing the required endovascular intervention at the time of procedure.
  The total sample size for this PMCF study is 100 patients, divided over up to 10 sites, throughout an enrolment period of 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Number of Patients without Serious Adverse Events (SAEs) and Serious Adverse Device Effects (SADEs | 30 days post procedure
  Primary Safety Endpoint
  Freedom from Serious Adverse Events (SAEs) and Serious Adverse Device Effects (SADEs)
Number of Patients without Serious Adverse Events (SAEs) and Serious Adverse Device Effects (SADEs | 30 days post procedure
  Primary Safety Endpoint
  Freedom from device and procedure related death.
Technical success rate | during surgery
  Technical success rate defined as successful crossing, introduction, deflation and a <30% residual stenosis on visual assessment of the SABER OTW PTA Catheter, SABERX PTA Catheter, and/or the Powerflex Pro PTA Catheter according to the respective IFU.
Number of Participants without Freedom from clinically-driven target lesion revascularization (CD-TLR) | 30 days post procedure
  Primary Efficacy Endpoint
  The primary efficacy endpoint is freedom from clinically-driven target lesion revascularization (CD-TLR)

SECONDARY OUTCOMES:
Technical success rate | during surgery
  Secondary Performance Endpoint
  Technical success rate defined as successful crossing, introduction, deployment and successful completion of the procedure of the Cordis guidewires (Emerald, ATW, Stablizer, Storq, SV 0.018", Wizdom) and/or the Cordis guiding catheters (Adroit, Vista Brite Tip) and/or the Cordis diagnostic catheters (Super Torque, Super Torque MB, Super Torque Plus, Infiniti 4F/5F/6F, Tempo 4F, Tempo Aqua, High Flow, Pigtail Straightener) and/or the Cordis vascular access devices (Avanti+, Brite Tip, Vista Brite IG, vessel dilator) and/or the Cordis vascular closure devices (MynxGrip and Mynx Control) and/or the Cordis OUTBACK CTO catheters according to the respective IFU.
Technical success rate | during surgery up to 24 hours after surgery
  Secondary Performance Endpoint
  Technical success rate defined as successful hemostasis without conversion to manual/mechanical compression of the Cordis vascular closure devices (MynxGrip and Mynx Control)
Number of Participants without Freedom from clinically-driven target lesion revascularization (CD-TLR) | 30 days post-procedure
  Secondary Performance Endpoint
  Freedom from clinically-driven target lesion revascularization (CD-TLR), defined as any reintervention at the target lesion due to symptoms
Change of ABI Index | 30 days post-procedure
  Secondary Performance Endpoint
  Change of Ankle Brachial Index (ABI), compared to baseline ABI
Time-to-hemostasis (HTC) | up to 24 hours after surgery
  Secondary Performance Endpoint
  Time-to-hemostasis assessed for the Cordis vascular closure devices (MynxGrip and Mynx Control). Categorized as Hemostatic time category (HTC) ≤2, HTC >2 to ≤4, HTC >4 to ≤5, HTC >5 to ≤7, HTC >7 to ≤10 min.
Time-to-ambulation | up to 24 hours after surgery
  Secondary Performance Endpoint
  Time-to-ambulation assessed for the Cordis vascular closure devices (MynxGrip and Mynx Control) defined as time between end of the procedure and ambulation in hours
Rate of Major Amputation free survival | 30 days post-procedure
  Secondary Safety Endpoint
  Rate of Major Amputation free survival defined as any amputation below the knee
Clinical success | 30 days post-procedure
  Secondary Safety Endpoint
  Clinical success, defined as an improvement of the Rutherford Classification of one class or more, as compared to the baseline Rutherford Classification (Rutherford Classification category from 0 to 6)
Number of Participants without Vessel perforation/dissection | during surgery
  Secondary Safety Endpoint
  Vessel perforation/dissection
Freedom from Serious Adverse Events | 30 days post-procedure
  Secondary Safety Endpoint
  Freedom from Serious Adverse Events (SAEs) and Serious Adverse Device Events (SADEs)
All cause of death | Through study completion
  Secondary Safety Endpoint
  All cause of death

CONTACTS AND LOCATIONS:
Locations (5):
- Austria (3):
  - Tirol Kliniken GmbH, Innsbruck
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Medizinische Universität, Vienna
- Germany (2):
  - Krankenhäuser Landkreis Freudenstadt gGmbH, Freudenstadt
  - SRH Klinikum Karlsbad-Langensteinbach GmbH, Langensteinbach

IPD SHARING:
Plan to Share IPD: No